CLINICAL TRIAL: NCT06330181
Title: Virtual Walking Therapy for Neuropathic Pain Following Incomplete Spinal Cord Injury
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Texas A&M University (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); Immersive Experience Labs (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SC220178; HT9425-23-1-1019 (Other Grant/Funding Number: Department of Depense); SC220178 (Other Grant/Funding Number: Congressionally Directed Medical Research Programs)
Record Dates: First submitted 2024-03-19; First posted 2024-03-26 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-04

CONDITIONS: Spinal Cord Injuries; Neuropathic Pain
Keywords: Spinal Cord Diseases; Central Nervous System Diseases; Trauma, Nervous System; Peripheral Nervous System Diseases; Neuromuscular Diseases; Pain; Neurologic Manifestations; Spinal Cord Injuries; Neuralgia; Wounds and Injuries
MeSH Terms: conditions — Spinal Cord Injuries; Neuralgia; Spinal Cord Diseases; Central Nervous System Diseases; Trauma, Nervous System; Peripheral Nervous System Diseases; Neuromuscular Diseases; Pain; Neurologic Manifestations; Wounds and Injuries

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of two intervention arms. Both groups receive the same number of sessions, duration of sessions, and measures procured.
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual reality (VR) game 1 (Active Comparator): Participants will be asked to play a virtual reality game twice a day for 10 days.
  Interventions: Other: VR Game 1
- Virtual reality (VR) game 2 (Active Comparator): Participants will be asked to play a virtual reality game twice a day for 10 days.
  Interventions: Other: VR Game 2

INTERVENTIONS:
Other: VR Game 1 — Individuals playing VR game 1 will wear a head-mounted display to allow them to visualize virtual legs in the virtual environment. When wearing the display, individuals will see the legs and arms of their virtual avatar from a first-person perspective.
  Individuals will engage in virtual reality sessions in their home twice daily over the course of 10 days in a two-week period. Each daily session will take approximately 30 minutes, with 5-10 minutes dedicated to the virtual walking experience. Additionally, each daily session will be scheduled a minimum of 4 hours apart
  Arms: Virtual reality (VR) game 1
Other: VR Game 2 — Individuals playing VR game 2 will wear a head-mounted display to allow them to visualize virtual legs in the virtual environment. When wearing the display, individuals will see the legs and arms of their virtual avatar from a first-person perspective.
  Individuals will engage in virtual reality sessions in their home twice daily over the course of 10 days in a two-week period. Each daily session will take approximately 30 minutes, with 5-10 minutes dedicated to the virtual walking experience. Additionally, each daily session will be scheduled a minimum of 4 hours apart.
  Arms: Virtual reality (VR) game 2

SUMMARY:
The purpose of this study is to determine if playing a virtual reality walking game can help improve neuropathic pain in adults with incomplete spinal cord injury.

DETAILED DESCRIPTION:
Many people with SCI experience neuropathic pain. Neuropathic pain is often described as sharp, burning, or electric. 'Traditional' treatments often do not do a good job of reducing neuropathic pain. Therefore, it is important to see if 'non-traditional' treatments might work. Scientists think that neuropathic pain occurs in SCI because the sensations coming from the eyes and up the spinal cord to the brain do not match what the brain thinks it told the body to do. This 'mismatch' may result in changes in the brain that make neuropathic pain possible. Virtual reality walking may potentially reduce this 'mismatch' by creating the 'illusion' that the person is walking. The brain then thinks it is telling the body to walk AND the information coming from the eyes matches its instructions. This 'matching' may reverse the brain changes that make neuropathic pain possible. The current study is specifically focused on individuals whose SCI has been classified as incomplete (ASIA B, C, or D).

ELIGIBILITY:
Inclusion Criteria:

The study will recruit individuals with incomplete injury (American Spinal Injury Association [ASIA] classification B, C, or D) with lumbar, paraplegic, or low tetraplegic (C5-C7) injury. Additional criteria will include:

1. Must have persistent NP symptoms that are of daily severity of at least 4/10 for 3 or more months
2. Must endorse more than 2 items on a 7-item Spinal Cord Injury Pain Instrument, SCIPI
3. Must be 18 years of age or older
4. Must be more than one and a half years post-injury to begin study (can be screened at an earlier time for eligibility)
5. Must have mobile connectivity with usable service
6. Must be stable on pain medication for 1 or more months
7. Must be cleared on the VRWalk physical activity clearance scale
8. Must not have motion sickness that interferes with daily life
9. Must use a wheelchair at least 75% of the time

Exclusion Criteria:

1. Individuals with Injury levels between C1 and C4
2. Individuals under the age of 18
3. Individuals who were injured within the past year
4. Individuals who cannot comprehend spoken English
5. Individuals who are in prison
6. Individuals who are blind
7. Individuals who experience severe motion sickness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-12-02 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Change in Pain Intensity | Baseline - final follow up (up to 18 months)
  The Numeric Rating Scale (NRS) measures pain intensity via a 0-10 numeric rating scale 0-10 where 0 is no pain, and 10 is the worst pain imaginable.

SECONDARY OUTCOMES:
Change in Pain Quality | Baseline - final follow up (up to 18 months)
  The Neuropathic Pain Scale (NPS) assesses the distinct pain qualities, including sharpness, heat/cold, dullness, intensity, overall unpleasantness, and surface vs. deep pain. The NPS consists of 10 items. 0 equals 'No sensation' and 10 equals 'Worst sensation imaginable.' All the items are rated 0-10 scale, with a higher score indicative of more neuropathic pain for each type of respective pain.
Change in Pain Interference | Baseline - final follow up (up to 18 months)
  The International Spinal Cord Injury Pain Basic Data Set version 2.0 interference assesses the degree to which pain interferes with day-to-day activities, mood, and sleep. Items are scored on a 0-10 numeric rating scale, and scores are summed to yield an interference score ranging from 0 to 30. Higher scores indicate greater interference from pain.
Post treatment change | at follow up (up to 18 months)
  The Patient Global Impression of Change is a one item 7 point Likert item assessing improvement of the participants' overall status. A score of 1 is 'Very Much Improved', and a score of 7 is 'Very Much Worse.' Higher scores indicate less perceived improvement.
  Range of scores: 1-7
Change in mood | Baseline - final follow up (up to 18 months)
  Mood will be assessed using the Patient Health Questionnaire-9. Participants will be asked to rate how often they have been bothered by specific problems on a 4-point Likert scale, where 0 is 'Not at all,' and 3 is 'Nearly every day.' The items are summed to yield a score ranging from 0-27. Higher scores indicate worse mood.
Change in quality of life | Baseline - final follow up (up to 18 months)
  Quality of life is assessed by the Satisfaction with Life Scale. This is a 5 item survey. Response options are a 7-point Likert scale where 1 is 'Strongly disagree,' and 7 is 'Strongly agree'. Items may be assessed individually or by summing items.
  Range of scores: 5-35. Higher scores indicate more satisfaction in life
Neurological changes | Baseline - 6 months
  For eligible and interested participants, functional Magnetic Resonance Imaging (fMRI) will be used to observe neurological changes. Pre and post-study images will be compared by experienced researchers.

CONTACTS AND LOCATIONS:
Locations (1):
- Texas A&M University, College Station, Texas, United States